CLINICAL TRIAL: NCT01683786
Title: An Open Label, Randomized, Parallel Design Estimation Pilot Study to Compare the Effectiveness of 36 vs 48 Wks PegIntron Plus Ribavirin Treatment for HCV Patients Without Rapid Virologic Response(RVR) But With Undetectable HCV RNA at wk 8
Brief Title: 36 vs 48 Wks Peg-Intron Plus Ribavirin for HCV Patients Without Rapid Virologic Response But Without HCV RNA at wk 8
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP39068
Record Dates: First submitted 2012-01-31; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegintron + Riba for 36 wks in total (Experimental): Pegylated IFN-α2b at 1.5 µg/kg of body weight/week and ribavirin 800~1400 mg/day for 24 weeks (36 weeks in total HCV treatment)
  Interventions: Drug: Pegintron + Riba
- Pegintron + Riba for 48 wks in total (Active Comparator): Pegylated IFN-α2b at 1.5 µg/kg of body weight/week and ribavirin 800~1400 mg/day for 36 weeks (48 weeks in total HCV treatment)
  Interventions: Drug: Pegintron + Riba

INTERVENTIONS:
Drug: Pegintron + Riba — Pegylated IFN-α2b at 1.5 µg/kg of body weight/week and ribavirin 800~1400 mg/day

SUMMARY:
Purpose:

To compare the effectiveness of 36 weeks versus 48 weeks pegintron plus ribavirin treatment for hepatitis C virus(HCV) patients without rapid virologic response(RVR), but with undetectable HCV RNA at wk 8.

Study Design:

a multi-site, prospective, open label, randomized, pilot trial. Approximately 60 HCV Genotype 1 patients who fail to achieve RVR but achieve undetectable HCV RNA at week 8 (<50 IU/ml) will be recruited into 2 arms(30 in each arm). Patients must receive pegylated interferon-α2b at 1.5 μg/kg of body weight/week and ribavirin 800~1400 mg/day for 12 wks before entering this study.

DETAILED DESCRIPTION:
Purpose:

To compare the effectiveness of 36 wks versus 48 wks pegintron plus ribavirin treatment for HCV patients without RVR, but with undetectable HCV RNA at wk 8.

Study Design:

This is a multi-site, prospective, open label, randomized, pilot trial. Approximately 60 HCV Genotype 1 patients who fail to achieve RVR at wk 4 but achieve undetectable HCV RNA at wk 8 (<50 IU/ml) will be recruited into 2 arms(30 in each arm). Patients must receive pegylated IFN-α2b at 1.5 μg/kg of body weight/week and ribavirin 800~1400 mg/day for 12 wks before entering this study.

Study Duration:

The estimated recruitment period is 12 months; the follow-up duration is 72 weeks (longest treatment period plus 6 month- f/u period); the total study duration (FPE->LPLV) is estimated to be 2.5 years

Statistical Analysis and Sample Size Justification:

A. The study is not primarily designed for hypothesis testing; thus the sample size calculation is not based on the primary objective, Approximately 60 subjects (30 in each arm) will be recruited into this study B. For descriptive statistics, the continuous variables will be expressed as mean ± standard deviation, and the categorical variables will be performed the number of cases and the corresponding percentages.

The primary analysis will focus on the efficacy response to the shortened HCV treatment course (36 wks) compared with standard course (48 wks). The between-group difference for efficacy endpoint will be assessed by the difference in the percentage of virologic responder after 24 wks of HCV treatment. For univariate analyses, comparisons of independent samples (shortened vs. standard course) will be assessed with Student's t test. The comparisons of categorical variables will be assessed using the chi-square test. Regarding the multivariate analysis, the proportion of patients achieving virologic responder will be compared among groups using a logistic regression analysis with terms of potential confounding factors. The OR estimates will be derived from the logistic regression model and the corresponding 95% CIs will be used to quantify the each effect of treatment course length and confounding factors.

All randomized patients who take at least one dose of HCV regimen will be included in safety assessment. Fisher's exact test will be used to compare between-group incidences of AEs. For patients with any clinical AEs, treatment related AEs, serious AEs, or discontinuations because of AEs, the data among groups will be provided as well. Statistical significance will be determined at the 0.05 level for all tests.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20y/o or older
2. Positive for the HCV antibody and HCV RNA detected with abnormal ALT (≧ 1X) before initiating PegIFN plus RBV treatment
3. HCV Genotype 1
4. Have failed to achieve RVR at week 4 but achieve undetectable HCV RNA at week 8 (< 50 IU/ml) with PegIFN plus RBV treatment
5. Have received PegIFN plus RBV treatment for 12weeks with good compliance (who have received >80% of expected PegIFN and RBV doses and completed at least 80% of the expected duration (80/80/80 adherence) and achieve EVR before entering this study

Exclusion Criteria:

1. Subjects with decompensated liver disease or overt cirrhosis by ultrasound.
2. With prior exposures to interferon (standard or pegylated) treatment before baseline.
3. With human immunodeficiency virus
4. With hepatitis B infection
5. With neutrophil count < 1500 mm3,
6. With platelet count < 90000 mm3,
7. With hemoglobin level < 12g/dL for men or < 11 g/dL for women
8. With serum creatinine level > 1.5 mg/dL
9. With clinically significant cardiac or cardiovascular abnormalities, organ grafts, systemic infections, clinically significant bleeding disorders, evidence of malignant neoplastic diseases
10. Female patients with pregnancy or lactation. Pregnancy in partners of male patients.
11. Hypersensitive to study drugs cases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The rate of sustained virologic response | At 24 weeks after end of treatment
  The comparison of the rates of sustained virologic response (SVR) defined as the proportion of patients with loss of serum HCV RNA at week 24 of post-treatment between patient groups (36 vs 48 weeks of treatment period)

SECONDARY OUTCOMES:
the factors associated with sustained virologic response(SVR) between groups | 24 weeks after the end of treatment
  the SVR assessment is defined as 24 weeks after the end of treatment, which mean 48 weeks after randomization for the shorten treatment arm and 60 weeks after randomization for the standard treatment arm
the rate of end-of-treatment response(EOT) | At the end of treatment (36 or 48 weeks of treatment period)
  The comparison of the rates of end-of-treatment response (EOT) defined as the proportion of patients with loss of serum HCV RNA at the end of treatment between patient groups (36 vs 48 weeks of treatment period)
The relapse rate | At 24 weeks after end of treatment
  The comparison of the relapse rates defined as the proportion of patients without detectable serum HCV RNA at the end of treatment but with detectable HCV RNA at 24 weeks after end of treatment between patient groups (36 vs 48 weeks of treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hui Hu, M.D., Principal Investigator — Chang Gung Medical Foundation, Kaohsiung Branch
Locations (5):
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung Branch, Kaohsiung City
  - Pingtung Christian Hospital, Pingtung City
  - Chi Mei Medical Center - Liouying Branch, Tainan
  - Shin Kong Wu Ho-Su Memorial Hosipital, Taipei